CLINICAL TRIAL: NCT04013139
Title: Evaluation of the Relationship Between Cardiopulmonary Exercise Testing (CPET ) Abnormalities and Ca-P Status in CKD Stage3-5
Brief Title: Relationship Between Cardiopulmonary Exercise Testing and Ca-P in Chronic Kidney Disease (CKD)
Status: Completed | Type: Observational
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Principal Investigator, Shahid Beheshti University of Medical Sciences
Other Study IDs: SBMU2314
Record Dates: First submitted 2019-06-23; First posted 2019-07-09 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Ckd-Mbd
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD Stage 3: CKD patients with GFR between 30-60cc/min
  Interventions: Diagnostic Test: CPET
- CKD Stage 4: CKD Patients with GFR 15-30 cc/min
  Interventions: Diagnostic Test: CPET

INTERVENTIONS:
Diagnostic Test: CPET — CPET

SUMMARY:
Reductions in exercise capacity associated with exercise intolerance augment cardiovascular disease risk and predict mortality in chronic kidney disease. This study utilized cardiopulmonary exercise testing to (a) investigate mechanisms of exercise intolerance; (b) unmask subclinical ca and p and vitamin D abnormalities that may precede cardiovascular disease in chronic kidney disease.

DETAILED DESCRIPTION:
Cardiopulmonary exercise testing will carry out in Stage 3-5 chronic kidney disease patients ; estimated glomerular filtration rate <60 ml/min/1.73 m2) and biochemistry will be added (Ca P Via D PTH FGF23).

ELIGIBILITY:
Inclusion Criteria:

* CKD Patients with GFR <60 non-dialysis
* age<18

Exclusion Criteria:

* HTN
* not signing consent
* active coronary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All >18 years CKD Patients with GFR <60 non-dialysis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Calcium x phosphorus change in stage 3-5 | 12 MONTHS
  CaxP change
CPET score change | 12 MONTHS
  Evaluation of CPET score change

SECONDARY OUTCOMES:
Renal Function change | 12 MONTHS
  GFR change

CONTACTS AND LOCATIONS:
Overall Officials: Dalili, Principal Investigator — SBMU
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No